CLINICAL TRIAL: NCT06110442
Title: Opportunistic Fragility Fracture Risk Estimates From Radiographs
Acronym: OFFER2
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 326406
Record Dates: First submitted 2023-09-20; First posted 2023-10-31 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: IbexBH Software — A software application applied to radiographs

SUMMARY:
The proposed study will predict a patients' risk of having osteoporosis by using a combination of the IBEX BH (Bone Health) software outputs and other clinical risk factors such as age, gender, medical history and lifestyle. A comparison will be made between the IBEX BH prediction and the one calculated in current clinical practice using a tool called FRAX (Fracture Risk Assessment Tool) which combines clinical risk factors with results from a Dual Energy X-ray Absorptiometry (DXA) assessment.

The study involves conducting these assessments on several new anatomies including Knee, Ankle and Pelvis, to extend the market reach and clinical utility of IBEX BH. The expected outcome of the study is that the IBEX BH will offer better decision support to clinicians in terms of referral on for a DXA scan or osteoporosis investigations than available today.

ELIGIBILITY:
For the collection of test data in the study.

Inclusion Criteria:

* Male or female
* 50 years of age or over

Exclusion Criteria:

* Women who are pregnant or are breastfeeding.
* Participants who have sustained fractures in both hips.
* Unwilling or unable to provide informed consent.

For the collection of healthy-normal data in the study.

Inclusion Criteria:

* Male or female
* 20-30 years of age

Exclusion Criteria:

* Women who are pregnant or are breastfeeding.
* Participants who have sustained fractures in both hips.
* Unwilling or unable to provide informed consent.

Ages: 20 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Representative population
Sampling Method: Non-Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
T-scores as calculated by IbexBH and DXA | 2 hours on 1 visit only

SECONDARY OUTCOMES:
Estimated 10-year risk of major osteoporotic fracture as outputted by FRAX (with and without DXA aBMD (Areal Bone Mineral Density) and IbexBH) | 2 hours on same visit as above

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No